CLINICAL TRIAL: NCT05828030
Title: Noninvasive Ventilation With High Flow Nasal Cannula Compared With Facial Mask in Patients With Chest Trauma: a Randomized Controlled Study
Brief Title: HFNC Compared With Facial Mask in Patients With Chest Trauma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202211029DIND
Record Dates: First submitted 2023-04-03; First posted 2023-04-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Chest Trauma; Hypoxia
MeSH Terms: conditions — Thoracic Injuries; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high flow nasal cannula group (Experimental): All patients will have FiO2 started at 0.4 and titrated to maintain oxygen saturation (SpO2) ≥ 95%. The flow rate will be set at titrated from 60 L/min.
  Interventions: Procedure: high flow nasal cannula
- Oxygen Mask group (Active Comparator): All patients will have FiO2 started at 0.4 and titrated to maintain oxygen saturation (SpO2) ≥ 95%.
  Interventions: Procedure: Oxygen mask

INTERVENTIONS:
Procedure: high flow nasal cannula — the patient receives HFNC after randomization. All patients will have FiO2 started at 0.4 and titrated to maintain oxygen saturation (SpO2) ≥ 95%.
  Arms: high flow nasal cannula group
Procedure: Oxygen mask — All patients will have FiO2 started at 0.4 and titrated to maintain oxygen saturation (SpO2) ≥ 95%.
  Arms: Oxygen Mask group

SUMMARY:
Guidelines for noninvasive ventilation (NIV) recommend continuous positive airway pressure in patients with thoracic trauma who remain hypoxic . However, no any suggestion was applied for high flow nasal cannula (HFNC). Therefore, Our aim was to determine whether HFNC reduces intubation in severe trauma-related hypoxemia.

DETAILED DESCRIPTION:
This would be a three-center randomized clinical trial of a level I trauma hospital. Inclusion criteria were patients with Arterial oxygen level (Pao2/)fraction of inspired oxygen inspired oxygen fraction(Fio2)<300 while receiving oxygen by high-flow mask within the first 72 h after thoracic trauma. Patients were randomized to remain on high-flow oxygen mask/ noninvasive ventilation or to receive HFNC. The interface was selected based on the associated injuries.

ELIGIBILITY:
Inclusion Criteria:

Patients who have the following condition within 72 hours of chest trauma despite receiving standard nasal cannula oxygen therapy [≥10 L/min], are eligible for inclusion.

* severe hypoxemic respiratory failure [Arterial partial pressure of oxygen (PaO2)/fraction of inspired oxygen fraction(FiO2) <300 mmHg]
* with a respiratory rate >25 breaths/minute and difficulty breathing, or respiratory distress
* PaCO2 of 45 mmHg or higher (if the patient requires emergency surgery with endotracheal intubation and mechanical ventilation, the time of inclusion will be the start of the post-extubation period. (Note: For patients who receive emergency trauma surgery with endotracheal intubation and mechanical ventilation, the time of inclusion assessment will be 72 hours after extubation.)

Exclusion Criteria:

1. Patients with a Glasgow Coma Scale less than 8 or severe brain injury.
2. Patients with any contraindications to non-invasive ventilation, including acute gastrointestinal bleeding, upper airway obstruction, or hemodynamic instability.
3. Facial trauma involving skull base fractures, facial bone fractures, or orbital floor fractures.
4. Severe injuries involving the nasal sinuses.
5. Patients with cervical spine injuries.
6. Patients with increased intracranial pressure.
7. Patients with facial, nasal, or airway structural abnormalities or surgery that prevents the use of appropriate nasal cannula.
8. Patients after upper airway surgery.
9. Patients who are unable to clearly express their willingness to sign informed consent.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of event of intubation or pneumonia | 30 days after randomization
  Intubation criteria included a respiratory rate of >40 breaths per minute, signs of increased breathing effort, SpO2 of <90% despite high fraction of inspired oxygen inspired oxygen fraction or acidosis with the quantitative measure of the acidity or basicity of aqueous or other liquid solutions (pH scale) of <7.35, occurrence of hemodynamic instability or deterioration of neurologic status.

SECONDARY OUTCOMES:
P/F ratio | 48 hrs after randomization
  P/F ratio would be count at the time 0/4/12/24/48 hours after randomization
pneumonia rate /tracheostomy rate | 30 days after randomization
  diagnosis of pneumonia was determined according to radiologic evidence of new or progressive infiltrate of more than 48 hours and laboratory detection of a causative agent.
  The management and diagnosis of all patients was performed by a trauma specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Chi Liao, MD, Principal Investigator — department of trauma of National University Hospital
Locations (2):
- Taiwan (2):
  - Department of Traumatology, National Taiwain University Hospital, Taipei, Taipei
  - NTUH Hsin-Chu Branch; NTUH Yun-Lin Branch, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No